CLINICAL TRIAL: NCT02978378
Title: Renal Biomarkers to Predict Recovery Following Venoarterial Extracorporeal Membrane Oxygenation
Status: Terminated | Type: Observational
Why Stopped: insufficient patients to satisfy study protocol(s) inclusion criteria
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Bonavia, Assistant Professor, Penn State Health Milton S Hershey Medical Center
Other Study IDs: STUDY00006088
Record Dates: First submitted 2016-11-17; First posted 2016-11-30 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2018-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and blood samples
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: biomarker levels — The level of the biomarker hyaluronic acid will be measured

SUMMARY:
The investigators objective is to assess the utility of renal biomarkers in predicting renal recovery following institution of Venoarterial Extracorporeal Membrane Oxygenation (VA-ECMO). Tissue biomarkers of renal injury may provide a real-time indication of renal function and the likelihood of renal recovery in patients having cardiogenic shock and requiring VA-ECMO. In these patients, traditional markers of kidney function (urine output and serum Creatinine level) do not accurately represent renal function.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* refractory or advanced cardiogenic shock prior to institution of VA-ECMO

Exclusion Criteria:

* History of chronic kidney disease prior to cardiogenic shock, as defined by estimated glomerular filtration rate (GFR) less than 60 mL per min
* Cognitive impairment
* Pregnant women
* patient or surrogate is not fluent in English
* Long-term immunosuppression

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cardiogenic shock and acute kidney injury requiring continuous renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
renal biomarker levels | through VA-ECMO decannulation, an average of 3 weeks
need for continuous renal replacement therapy at hospital discharge (Yes/No) | measured at hospital discharge, an average of 2-3 months following initial hospital admission
  The need for continuous renal replacement therapy at hospital discharge will be assessed using hospital medical records

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bonavia, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided